CLINICAL TRIAL: NCT05979233
Title: One Session Vs Staged Laropendoscopic Management of Calcular Obstructive Jaundice
Brief Title: One Session Vs Staged Management of Calcular Obstructive Jaundice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, MD, professor & consultant of general surgery, Department of surgery, Minia university hospital, Egypt, Minia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fac.med.23.42
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Calcular Obstructive Jaundice; Gall Bladder Disease
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- staged managment (Active Comparator): ERCP then interval laparoscopic cholecystectomy
  Interventions: Procedure: staged managment
- one session ERCP then LC (Experimental): one session ERCP then LC
  Interventions: Procedure: one session ERCP then LC
- one session LC then ERCP (Experimental): one session LC then ERCP
  Interventions: Procedure: one session LC then ERCP

INTERVENTIONS:
Procedure: staged managment — staged management
  Arms: staged managment
Procedure: one session ERCP then LC — one session ERCP then LC
  Arms: one session ERCP then LC
Procedure: one session LC then ERCP — one session LC then ERCP
  Arms: one session LC then ERCP

SUMMARY:
to compare the outcomes between doing ERCP and laparoscopic cholecystectomy in one session Vs staged management

DETAILED DESCRIPTION:
to compare the outcomes between 3 groups: in the 1st group we will do ERCP then laparoscopic cholecystectomy in the same session, in the 2nd group we will do laparoscopic cholecystectomy then ERCP in the same session in group 3 we will do staged management

ELIGIBILITY:
Inclusion Criteria:

* age from 18-70 year
* combined CBD and gall stone
* stone less than 1.5 cm
* fit for surgery
* no upper abdominal surgery

Exclusion Criteria:

* age <18 and >70
* unfit for surgery
* stone more than 1.5 cm
* upper abdominal surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-08-05 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
total cost | 6 months
  total cost in Egyptian pound
hospital stay | 6 months
  total hospital stay in days

SECONDARY OUTCOMES:
complications | 30 days
  early postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Minya, Egypt